CLINICAL TRIAL: NCT05197452
Title: Alive Church Network: Increasing COVID-19 Testing in Chicago's African American Testing Deserts
Brief Title: Increasing COVID-19 Testing in Chicago's African American Testing Desserts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20110407; R01NR018463 (NIH)
Record Dates: First submitted 2022-01-13; First posted 2022-01-19 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Testing

STUDY DESIGN:
Intervention Model Description: We established a network of testing sites in African American churches and community sites located in testing deserts in Chicago. Individuals of all ages were eligible for testing. Individuals with a confirmed COVID-19 infection within the past 3 months were ineligible. Testing was open to the public and no appointments were necessary. Testing was offered 5 days per week (at 1 or 2 locations each day) with varying hours of operation to accommodate community member's work and school schedules. There was no limit to the number of times an individual could be tested.
  Testing was administered by experienced mobile clinical teams of community health workers and registered nurses from Rush University Medical Center. Participants received COVID-19 education, social determinants of health screening, and free SARS-CoV-2 polymerase chain reaction (PCR) testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Testing (Experimental): COVID-19 antigen and PCR Testing
  Interventions: Behavioral: COVID-19 Testing

INTERVENTIONS:
Behavioral: COVID-19 Testing — For in-person PCR testing, a nasal swab will be inserted shallowly into the participant's nose and rotated in each nostril. The swab will be broken off into a designated test tube and placed into a specimen bag along with a label. All specimens will be stored in a cooler until they are transported the Rush Laboratory for COVID-19 analysis.
  For at home antigen testing, participants will download an app to their mobile phone and watch an informational video. The test will be self-administered by inserting a nasal swab into the nostril until a cap containing the swab touches the nose; rubbing the swab tip around the nose cavity 3 times; removing the swab and repeating in the other nostril. The nasal swab, a dropper, processing fluid, and a blue tooth connected analyzer are provided with the testing kit to analyze the sample for COVID-19. COVID-19 home test results are displayed on the participants smart phone after 15 minutes.

SUMMARY:
This study uses a population-based approach to increase uptake of COVID-19 testing within a highly segregated and underserved African American community in Chicago.

DETAILED DESCRIPTION:
The epidemic of novel coronavirus disease 2019 (COVID-19) has caused an unprecedented public health crisis in the United States. African Americans (AA) have been disproportionately impacted, as systemic inequities have contributed to increased exposure and vulnerability to COVID-19. Evidence suggests that AAs are delaying testing and care for COVID-19, which increases risk of transmission and poor outcomes. In Chicago, segregated AA neighborhoods have experienced some of the highest COVID-19 mortality rates in the city, yet large portions of these neighborhoods remain testing deserts. Providing trusted, accessible, community-based testing in underserved AA communities is critical to ensuring that AAs receive an early diagnosis, thereby reducing the risk of further transmission and improving clinical outcomes. This study leverages the Alive Church Network (ACN), a long-standing, community-driven coalition of African American pastors and public health researchers that was developed as a sustainable infrastructure to address health inequities in chronic disease in segregated AA neighborhoods in Chicago. The ACN was designed to address lack of access to health care, cultural insensitivity, and lack of trust, which are the root cause of disparities in chronic disease as well as infectious disease, including COVID-19. This project utilizes the ACN infrastructure to create a network of church-based testing sites in a segregated and underserved AA neighborhood in Chicago that will provide COVID-19 testing and education as well as linkage to healthcare and social resources. Pastors who serve predominantly AA congregations on the South Side of Chicago will form a coalition to promote community-wide COVID-19 testing in local churches and church-based events where residents are congregating, such as Sunday church services, food pantries, and other gatherings. Residents of all ages will receive COVID-19 education and free severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction (PCR) testing with rapid turn-around of results from an on-site clinical team, as well as connection to local resources to address social needs, including food, housing, and medical care. At-home COVID-19 tests will also be provided to residents for their personal use and to distribute to others in their social network. The primary aim of the study is to evaluate the impact of the ACN COVID-19 testing intervention on uptake of testing among residents of target high poverty AA neighborhoods in Chicago.

ELIGIBILITY:
Inclusion Criteria:

• All individuals who request a COVID-19 test, including pregnant women and children of all ages

Exclusion Criteria:

• Individuals who have tested positive for Covid-19 in the prior 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2167 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lynch, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm Only: We only had a single arm in this trial because there were not sufficient data points to test our original hypothesis. The intervention arm consisted of individuals who received a Covid PCR test. Enrollment is closed and all collected data is currently reported.
Period: Overall Study
Arm/Group | Intervention Arm Only
Started | 2167
Completed (Enrollment closed. All collected data reported.) | 2167
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- COVID-19 Testing: COVID-19 antigen and PCR Testing
  COVID-19 Testing: For in-person PCR testing, a nasal swab will be inserted shallowly into the participant's nose and rotated in each nostril. The swab will be broken off into a designated test tube and placed into a specimen bag along with a label. All specimens will be stored in a cooler until they are transported the Rush Laboratory for COVID-19 analysis.
  For at home antigen testing, participants will download an app to their mobile phone and watch an informational video. The test will be self-administered by inserting a nasal swab into the nostril until a cap containing the swab touches the nose; rubbing the swab tip around the nose cavity 3 times; removing the swab and repeating in the other nostril. The nasal swab, a dropper, processing fluid, and a blue tooth connected analyzer are provided with the testing kit to analyze the sample for COVID-19. COVID-19 home test results are displayed on the participants smart phone after 15 minutes.
  At home testing was performed by inserting a nasal swab into the nostril until the cap containing the swab touched the nose; rubbing the swab tip around the nose cavity 3 times; removing the swab and repeating in the other nostril. The nasal swab, a dropper, processing fluid, and a blue tooth connected analyzer were provided with the testing kit to analyze the sample for Covid-19. Covid-19 home test results are displayed on the participants smart phone after 15 minutes.
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 2167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 264
  Between 18 and 65 years | 1582
  >=65 years | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1184
  Male | 983
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1506
  White | 152
  More than one race | 14
  Unknown or Not Reported | 489
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2167

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Testing Uptake
Description: Covid testing uptake was measured as the number of neighborhood residents (i.e., count of unique participants) tested for COVID-19 at any timepoint during the study which occurred between December 2020 and August 2022. The were 397 testing events at churches or community site where participants could be tested during this time period. Individuals may have been tested more than once but were only counted once. Testing uptake was assessed as the number of participants tested at least once (n=2167). Pre and post evaluations were not performed. The measure was based a single count of participants tested.
Time Frame: Up to 20 months
Population: The analysis population included unique individuals tested for Covid-19
Measure: Count of Participants; unit: Participants
Groups:
- COVID-19 Testing: COVID-19 antigen and PCR Testing
  COVID-19 Testing: For in-person PCR testing, a nasal swab will be inserted shallowly into the participant's nose and rotated in each nostril. The swab will be broken off into a designated test tube and placed into a specimen bag along with a label. All specimens will be stored in a cooler until they are transported the Rush Laboratory for COVID-19 analysis.
  For at home antigen testing, participants will download an app to their mobile phone and watch an informational video. The test will be self-administered by inserting a nasal swab into the nostril until a cap containing the swab touches the nose; rubbing the swab tip around the nose cavity 3 times; removing the swab and repeating in the other nostril. The nasal swab, a dropper, processing fluid, and a blue tooth connected analyzer are provided with the testing kit to analyze the sample for COVID-19. COVID-19 home test results are displayed on the participants smart phone after 15 minutes.
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 2167
Participants | 2167

2. Other Pre Specified Outcome: Re-AIM Framework
Description: Use the RE-AIM framework to assess the Reach, Effectiveness, Adoption, Implementation, and Maintenance of the ACN COVID-19 testing intervention.
Time Frame: Up to 6 months after end of study
Population: We did not have enough enrolled participants to assess this outcome.
Groups:
- Intervention Arm Only: We only had a single arm in this trial because there were not sufficient data points to test our original hypothesis. The intervention arm consisted of individuals who received a Covid PCR test.
Arm/Group | Intervention Arm Only
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Needs Assessment
Description: Evaluate COVID-19 testing history, attitudes towards COVID-19 testing, and perceived risk of COVID-19 via survey.
Time Frame: First 2 months of the study prior to the start of the testing intervention
Population: 215 participants who completed the needs assessment survey
Measure: Number; unit: participants
Groups:
- Needs Assessment: Of 955 participants of a previous health screening in the target neighborhood, 394 (41.3%) were contacted and 215 (22.5%) agreed to participate in the COVID-19 needs assessment survey.
Arm/Group | Needs Assessment
Number analyzed (Participants) | 215
participants
  Tested for Covid-19 at least once | 112
  Previously tested positive for Covid-19 | 20
  Had a family member, friend, or colleague who tested positive for Covid 19 | 183
  Had a family member, friend, or colleague who died from Covid 19 | 129
  Thought a family member, friend or colleague would get Covid 19 in the future | 185
  Thought that they themselves would get Covid 19 in the future | 90
  Would get tested at a church in their neighborhood if availble | 182

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: Staff members recorded any adverse events that occurred during testing. We did not monitor adverse events after testing since this not was not a part of our intervention (i.e., there was no designated follow-up period). There were no adverse or serious adverse events reported.
Arm/Group | Intervention Arm Only
All-Cause Mortality (participants affected / at risk) | 0/2167
Serious Adverse Events (participants affected / at risk) | 0/2167
Other Adverse Events (participants affected / at risk) | 0/2167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT05197452/Prot_000.pdf